CLINICAL TRIAL: NCT00255762
Title: Phase II Trial of Carboplatin, Weekly Paclitaxel and Biweekly Bevacizumab in Patients With Unresectable Stage IV Melanoma
Brief Title: Carboplatin, Paclitaxel, and Bevacizumab in Treating Patients With Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01823; NCI-2012-01823 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000449967; NCCTG-N047A (Other: North Central Cancer Treatment Group); N047A (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Carboplatin; Paclitaxel; Taxes; Bevacizumab

ARMS (1):
- Treatment (carboplatin, paclitaxel, bevacizumab) (Experimental): Patients receive carboplatin IV over 30 minutes on day 1, paclitaxel IV over 1 hour on days 1, 8, and 15, and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving carboplatin and paclitaxel together with bevacizumab works in treating patients with stage IV melanoma that cannot be removed by surgery. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving carboplatin and paclitaxel together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the anti-tumor activity of carboplatin, paclitaxel, and bevacizumab, in terms of progression-free survival, in patients with unresectable stage IV melanoma.

II. Determine the toxicity profile of this regimen in these patients.

Secondary I. Determine the distribution of overall survival times in patients treated with this regimen.

II. Determine the response rate in patients treated with this regimen. III. Determine the changes in blood levels of vascular endothelial growth factor in patients treated with this regimen.

IV. Determine the changes in immune homeostasis in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV over 30 minutes on day 1, paclitaxel IV over 1 hour on days 1, 8, and 15, and bevacizumab IV over 30-90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 47 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma

  * Unresectable stage IV disease
  * Evidence of metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No radiologically confirmed invasion of adjacent organs (e.g., duodenum or stomach)
* No tumor invasion of major blood vessels
* No history of primary brain tumor or other CNS disease
* No brain metastases by MRI or CT scan
* Performance status - ECOG 0-2
* More than 4 months
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion allowed)
* No active bleeding
* Bilirubin ≤ 1.5 mg/dL
* AST ≤ 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* INR ≤ 1.5 times ULN
* PTT normal
* No known esophageal varices
* Creatinine ≤ 1.5 times ULN
* Urine protein creatinine ratio ≤ 0.5
* Urine protein < 1 g/24-hr urine collection
* No New York Heart Association class II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No myocardial infarction within the past 6 months
* No unstable angina within the past 6 months
* No clinically significant peripheral vascular disease
* No uncontrolled hypertension (i.e., blood pressure ≥ 150/90 mmHg despite antihypertensive therapy)
* No clinically significant stroke within the past 6 months
* No deep vein thrombosis within the past year
* No other vascular abnormality
* No pulmonary embolus within the past year
* No history of abdominal fistula
* No gastrointestinal perforation
* No intra-abdominal abscess within the past 4 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* No other pathological condition that would confer a high risk of bleeding
* No active infection requiring parenteral antibiotics
* No serious nonhealing wound (including wounds healing by secondary intention), ulcer, or bone fracture
* No peripheral neuropathy ≥ grade 2
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to the study drugs
* No uncontrolled seizures
* No other uncontrolled illness
* No significant traumatic injury within the past 4 weeks
* No prior antivascular endothelial growth factors (VEGF), including any of the following:

  * Bevacizumab
  * VEGF Trap
  * Anti-VEGF receptor monoclonal antibody
  * Small molecular tyrosine kinase inhibitors of VEGF receptors
* No more than 1 prior systemic chemotherapy regimen
* No prior carboplatin or paclitaxel
* No other concurrent chemotherapy
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25% of bone marrow
* No concurrent radiotherapy
* At least 4 weeks since prior major surgical procedure or open biopsy
* At least 1 week since prior fine-needle aspiration or core biopsy
* No concurrent major surgery
* More than 4 weeks since prior systemic therapy
* No concurrent full-dose oral or parenteral anticoagulation

  * No concurrent antiplatelet therapy except low-dose aspirin (i.e., 81 mg of oral aspirin daily) allowed
* No other concurrent experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Time from registration to documentation of disease progression, assessed up to 8 weeks
  Constructed using the properties of the binomial distribution. Estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Confirmed tumor response (complete response or partial response) | Up to 5 years
  A ninety percent confidence interval for the true proportion of confirmed tumor responses will be calculated assuming that the number of confirmed tumor responses follows a binomial distribution.
Clinical response rate | Up to 5 years
  A ninety percent confidence interval for the true clinical response rate will be calculated.
Overall survival | Time is defined as the time from registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States